CLINICAL TRIAL: NCT02831296
Title: Prospective Evaluation of Infants With Spinal Muscular Atrophy: SPOT SMA
Brief Title: Prospective Evaluation of Infants With Spinal Muscular Atrophy:
Acronym: SPOTSMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Utah (Other); University of Massachusetts, Worcester (Other); ARUP Laboratories (Other); Newborn Screening Translational Research Network (Unknown); American College of Medical Genetics and Genomics (Unknown); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Kathryn J Swoboda, Katherine B. Sims MD Endowed Chair in Neurogenetics, Massachusetts General Hospital
Other Study IDs: 2015P001934; R01HD069045 (NIH)
Record Dates: First submitted 2016-07-01; First posted 2016-07-13 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Spinal Muscular Atrophy
Keywords: SMA; Werdnig-Hoffmann disease; Kugelberg-Welander disease
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — DNA, RNA and specific biomarker assessments for whole blood SMN protein levels, plasma and serum for exploratory metabolomics profiling, skin biopsy for fibroblast cell line establishment (iPS cell line studies)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Affected Subjects <36 Mos. of Age: Infants and children 36 months of age and younger at time of enrollment who have been genetically diagnosed with Spinal Muscular Atrophy (SMA)
  The affected cohort will receive coordinated, multidisciplinary care including dietary intervention, respiratory monitoring, physical therapy, and genetic counseling. They will also undergo assessment of motor function, muscle action potential measurement, and body composition, as well as blood sample collection for DNA and biomarkers, and optional research skin biopsy.
- Unaffected Subjects <36 Mos. of Age: Infants and children 36 months of age and younger who are not affected with SMA
  The unaffected group will undergo the same assessments as the affected group.
- Unaffected Family Members: Parents and siblings of any age, without genetic diagnosis of SMA, who have family members enrolled in either of the Affected Infants/Children/Adults cohorts.
  The unaffected siblings will undergo the same assessments as the affected group, where age-appropriate. Unaffected parents' participation will be limited to blood sample collection and optional research skin biopsy.
- Affected Subjects >36 Mos. of Age: Children and adults >36 months at time of enrollment who have been genetically diagnosed with Spinal Muscular Atrophy.
  The older affected cohort will receive coordinated, multidisciplinary care including dietary intervention, respiratory monitoring, physical therapy, and genetic counseling. They will also undergo assessment of motor function, muscle action potential measurement, and body composition, as well as blood sample collection for DNA and biomarkers, and optional research skin biopsy. Where applicable, these participants will be considered Affected Control Subjects.

SUMMARY:
SPOT SMA is a prospective NIH-supported clinical study targeting pre-symptomatic or recently diagnosed infants and children with Spinal Muscular Atrophy (SMA) types 1, 2, or 3 and their healthy control siblings less than 36 months of age at the time of study enrollment. The main objective of the study is to prospectively collect longitudinal clinical outcomes and provide counseling and education to parents of newly diagnosed children. The study will assess the impact of current standard of care management paradigms and interventions on health outcomes in newly diagnosed SMA infants and children with type 1, 2 or 3 and age appropriate controls. There is no investigational drug and no specific intervention in this study. Rather, the investigators will document outcomes related to current therapies provided to participating subjects, and will educate participants about possible clinical trial opportunities.

DETAILED DESCRIPTION:
Overview of data to be collected from enrolled infants followed longitudinally and entered into the NBSTRN Longitudinal Pediatric Data Resource

1. Past medical history relevant to pregnancy, delivery, complications in the immediate neonatal period, birth parameters, family history and any medical problems other than SMA (ie prematurity, etc)
2. Ongoing medical history indicating problems related to the following areas:

   feeding, growth, respiratory status including use of cough assist and bilevel respiratory support, gastrointestinal issues, cardiac symptoms, neurologic symptoms or signs including muscle weakness, hospitalizations, ER visits, other adverse events
3. Assessment of dietary intake and use of nutritional supplements
4. Surgical history and ongoing documentation of assessments and need for g-tube, Nissen, tympanostomy, adenoidectomy/tonsillectomy or other airway surgeries, and orthopedic procedures
5. Caregiver obtained developmental history and documentation of newly acquired and/or loss of previously acquired gross motor skills at the time of each visit
6. Documentation of caregiver reported outcomes
7. Documentation of anthropometric measures, vital signs, general physical examination parameters
8. Neurological examination using standardized tools
9. Time to death, permanent invasive ventilation and/or need for > 16 hours/day of bilevel respiratory support
10. Specific assessment of motor function as measured using age appropriate motor outcome measures such as: the Children's Hospital of Philadelphia Infant Tests of Neuromuscular Disorders (CHOP-INTEND), Test of Infant Motor Performance Screening Inventory, WHO motor milestones or others, and Hammersmith Functional Motor Scale for SMA Expanded for children 18 months and older
11. Electrophysiologic studies such as maximum ulnar compound muscle action potential (CMAP) amplitude and area
12. Documentation of range of motion, development of limb contractures and/or presence of scoliosis, lordosis, hip dysplasia or other orthopedic outcomes
13. Additional optional exploratory biomarker assessments
14. DEXA measurements to assess body composition and bone density
15. The option to enroll in an autopsy study at the time of death to contribute samples to a research biorepository

Normal control subjects such as unaffected siblings will undergo these same measurements, as applicable. Unaffected parents' participation will be limited to collection and banking of blood and cell lines.

ELIGIBILITY:
Inclusion Criteria:

* For affected subjects: genetic diagnosis of SMA
* For unaffected family members: parent or sibling of any age (without genetic diagnosis of SMA) of affected subject enrolled in study

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pre-symptomatic or newly diagnosed infants and children with Spinal Muscular Atrophy (SMA) types 1, 2, or 3; OR unaffected parents and siblings of enrolled infants and children with SMA; OR control subjects: infants and children who are not affected with SMA
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-02; Primary Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Time to death and/or full time invasive ventilation or need for > 16 hours/day of bilevel respiratory support | At each visit (every 1-6 months depending on age)

SECONDARY OUTCOMES:
Maximum Ulnar CMAP Amplitude | At each visit (every 1-6 months depending on age)
  Maximum ulnar compound muscle action potential (CMAP) amplitude and area
CHOP-INTEND | At each visit (every 1-6 months depending on age, or until deemed no longer appropriate by PI/physical therapist)
  Assessment of motor function in infants and children functioning at an infant level
WHO Motor Milestones | At each visit (every 1-6 months depending on age)
  Acquisition of gross motor milestones, per WHO guidelines
Hammersmith Functional Motor Scale - Expanded | At each visit (every 1-6 months depending on age, beginning when deemed appropriate by PI/physical therapist)
  Assessment of motor function in subjects whose motor function exceeds that of an infant
Hammersmith Infant Neurological Exam (HINE) | At each visit (every 1-6 months depending on age, beginning when deemed appropriate by PI/physical therapist)
  Assessment of neuromotor function in infants, general neurologic exam in infants
Body composition | Every 6 months
  DEXA scans
Bone density | Every 6 months
  DEXA scans
Need for tube feeding | At each visit (every 1-6 months depending on age)
Caregiver Questionnaire total score and subscores | At each visit (every 1-3 months depending on age and SMA type)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn J Swoboda, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The National Institute of Child Health and Human Development has a contract with the American College of Medical Genomics and the Newborn Screening Translational Research Network (NBSTRN) in collaboration with the bioinformatics group at the Cincinnati Children's Hospital to develop a national database for data capture and management for all the follow-up data to be collected for those who agree to participate in the research study. The investigators will share deidentified data with the NBSTRN database.
  The investigators will also submit relevant associated data (e.g., phenotype data) to an NIH-designated data repository in a timely manner, as indicated by the NIH Genomic Data Sharing policy.
  Aggregate Data will be available for submission/general research use.
Supporting Information: CSR
URL: https://nbstrn.org/supported-projects/spinal-muscular-atrophy

REFERENCES:
- [Background] Bitton A, Martin C, Landon BE. A nationwide survey of patient centered medical home demonstration projects. J Gen Intern Med. 2010 Jun;25(6):584-92. doi: 10.1007/s11606-010-1262-8. PMID 20467907
- [Background] Butchbach ME, Rose FF Jr, Rhoades S, Marston J, McCrone JT, Sinnott R, Lorson CL. Effect of diet on the survival and phenotype of a mouse model for spinal muscular atrophy. Biochem Biophys Res Commun. 2010 Jan 1;391(1):835-40. doi: 10.1016/j.bbrc.2009.11.148. Epub 2009 Nov 27. PMID 19945425
- [Background] Butchbach ME, Singh J, Thorsteinsdottir M, Saieva L, Slominski E, Thurmond J, Andresson T, Zhang J, Edwards JD, Simard LR, Pellizzoni L, Jarecki J, Burghes AH, Gurney ME. Effects of 2,4-diaminoquinazoline derivatives on SMN expression and phenotype in a mouse model for spinal muscular atrophy. Hum Mol Genet. 2010 Feb 1;19(3):454-67. doi: 10.1093/hmg/ddp510. Epub 2009 Nov 6. PMID 19897588
- [Background] Chung BH, Wong VC, Ip P. Spinal muscular atrophy: survival pattern and functional status. Pediatrics. 2004 Nov;114(5):e548-53. doi: 10.1542/peds.2004-0668. Epub 2004 Oct 18. PMID 15492357
- [Background] Cobben JM, Lemmink HH, Snoeck I, Barth PA, van der Lee JH, de Visser M. Survival in SMA type I: a prospective analysis of 34 consecutive cases. Neuromuscul Disord. 2008 Jul;18(7):541-4. doi: 10.1016/j.nmd.2008.05.008. Epub 2008 Jun 24. PMID 18579378
- [Background] Lefebvre S, Burglen L, Reboullet S, Clermont O, Burlet P, Viollet L, Benichou B, Cruaud C, Millasseau P, Zeviani M, et al. Identification and characterization of a spinal muscular atrophy-determining gene. Cell. 1995 Jan 13;80(1):155-65. doi: 10.1016/0092-8674(95)90460-3. PMID 7813012
- [Background] Lemoine TJ, Swoboda KJ, Bratton SL, Holubkov R, Mundorff M, Srivastava R. Spinal muscular atrophy type 1: are proactive respiratory interventions associated with longer survival? Pediatr Crit Care Med. 2012 May;13(3):e161-5. doi: 10.1097/PCC.0b013e3182388ad1. PMID 22198810
- [Background] Lorson CL, Hahnen E, Androphy EJ, Wirth B. A single nucleotide in the SMN gene regulates splicing and is responsible for spinal muscular atrophy. Proc Natl Acad Sci U S A. 1999 May 25;96(11):6307-11. doi: 10.1073/pnas.96.11.6307. PMID 10339583
- [Background] Mailman MD, Heinz JW, Papp AC, Snyder PJ, Sedra MS, Wirth B, Burghes AH, Prior TW. Molecular analysis of spinal muscular atrophy and modification of the phenotype by SMN2. Genet Med. 2002 Jan-Feb;4(1):20-6. doi: 10.1097/00125817-200201000-00004. PMID 11839954
- [Background] Mannaa MM, Kalra M, Wong B, Cohen AP, Amin RS. Survival probabilities of patients with childhood spinal muscle atrophy. J Clin Neuromuscul Dis. 2009 Mar;10(3):85-9. doi: 10.1097/CND.0b013e318190310f. PMID 19258855
- [Background] Oskoui M, Levy G, Garland CJ, Gray JM, O'Hagen J, De Vivo DC, Kaufmann P. The changing natural history of spinal muscular atrophy type 1. Neurology. 2007 Nov 13;69(20):1931-6. doi: 10.1212/01.wnl.0000290830.40544.b9. PMID 17998484
- [Background] Rudnik-Schoneborn S, Berg C, Zerres K, Betzler C, Grimm T, Eggermann T, Eggermann K, Wirth R, Wirth B, Heller R. Genotype-phenotype studies in infantile spinal muscular atrophy (SMA) type I in Germany: implications for clinical trials and genetic counselling. Clin Genet. 2009 Aug;76(2):168-78. doi: 10.1111/j.1399-0004.2009.01200.x. PMID 19780763
- [Background] Stange KC, Nutting PA, Miller WL, Jaen CR, Crabtree BF, Flocke SA, Gill JM. Defining and measuring the patient-centered medical home. J Gen Intern Med. 2010 Jun;25(6):601-12. doi: 10.1007/s11606-010-1291-3. PMID 20467909
- [Background] Stille C, Turchi RM, Antonelli R, Cabana MD, Cheng TL, Laraque D, Perrin J; Academic Pediatric Association Task Force on Family-Centered Medical Home. The family-centered medical home: specific considerations for child health research and policy. Acad Pediatr. 2010 Jul-Aug;10(4):211-7. doi: 10.1016/j.acap.2010.05.002. No abstract available. PMID 20605546
- [Background] Swoboda KJ, Prior TW, Scott CB, McNaught TP, Wride MC, Reyna SP, Bromberg MB. Natural history of denervation in SMA: relation to age, SMN2 copy number, and function. Ann Neurol. 2005 May;57(5):704-12. doi: 10.1002/ana.20473. PMID 15852397
- [Background] Swoboda KJ, Kissel JT, Crawford TO, Bromberg MB, Acsadi G, D'Anjou G, Krosschell KJ, Reyna SP, Schroth MK, Scott CB, Simard LR. Perspectives on clinical trials in spinal muscular atrophy. J Child Neurol. 2007 Aug;22(8):957-66. doi: 10.1177/0883073807305665. PMID 17761650
- [Background] Swoboda KJ, Scott CB, Reyna SP, Prior TW, LaSalle B, Sorenson SL, Wood J, Acsadi G, Crawford TO, Kissel JT, Krosschell KJ, D'Anjou G, Bromberg MB, Schroth MK, Chan GM, Elsheikh B, Simard LR. Phase II open label study of valproic acid in spinal muscular atrophy. PLoS One. 2009;4(5):e5268. doi: 10.1371/journal.pone.0005268. Epub 2009 May 14. PMID 19440247
- [Background] Swoboda KJ. Seize the day: Newborn screening for SMA. Am J Med Genet A. 2010 Jul;152A(7):1605-7. doi: 10.1002/ajmg.a.33519. No abstract available. PMID 20583173
- [Background] Wan L, Battle DJ, Yong J, Gubitz AK, Kolb SJ, Wang J, Dreyfuss G. The survival of motor neurons protein determines the capacity for snRNP assembly: biochemical deficiency in spinal muscular atrophy. Mol Cell Biol. 2005 Jul;25(13):5543-51. doi: 10.1128/MCB.25.13.5543-5551.2005. PMID 15964810
- [Background] Wirth B, Brichta L, Schrank B, Lochmuller H, Blick S, Baasner A, Heller R. Mildly affected patients with spinal muscular atrophy are partially protected by an increased SMN2 copy number. Hum Genet. 2006 May;119(4):422-8. doi: 10.1007/s00439-006-0156-7. Epub 2006 Mar 1. PMID 16508748
- [Background] Zerres K, Rudnik-Schoneborn S. Natural history in proximal spinal muscular atrophy. Clinical analysis of 445 patients and suggestions for a modification of existing classifications. Arch Neurol. 1995 May;52(5):518-23. doi: 10.1001/archneur.1995.00540290108025. PMID 7733848
- [Background] Kolb SJ, Coffey CS, Yankey JW, Krosschell K, Arnold WD, Rutkove SB, Swoboda KJ, Reyna SP, Sakonju A, Darras BT, Shell R, Kuntz N, Castro D, Iannaccone ST, Parsons J, Connolly AM, Chiriboga CA, McDonald C, Burnette WB, Werner K, Thangarajh M, Shieh PB, Finanger E, Cudkowicz ME, McGovern MM, McNeil DE, Finkel R, Kaye E, Kingsley A, Renusch SR, McGovern VL, Wang X, Zaworski PG, Prior TW, Burghes AH, Bartlett A, Kissel JT; NeuroNEXT Clinical Trial Network and on behalf of the NN101 SMA Biomarker Investigators. Baseline results of the NeuroNEXT spinal muscular atrophy infant biomarker study. Ann Clin Transl Neurol. 2016 Jan 21;3(2):132-45. doi: 10.1002/acn3.283. eCollection 2016 Feb. PMID 26900585